CLINICAL TRIAL: NCT06047002
Title: Panther (Personalised Antiplatelet Therapy for Patients With Symptomatic Peripheral Arterial Disease)
Brief Title: Personalised Antiplatelet Therapy for Patients With Symptomatic Peripheral Arterial Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0829
Record Dates: First submitted 2023-09-06; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples are being stored for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Peripheral arterial disease (PAD) is a condition where the blood vessels in the legs get blocked. It affects one out of every five adults over the age of 65. As it is the main cause of amputations, the NHS performs over 20,000 operations every year to prevent them. People with PAD benefit from tablets to thin their blood as this improves outcomes after surgery and prevents heart attacks and strokes. The main tablets for this purpose are aspirin and clopidogrel. These work in most people, but up to a third of patients do not get any benefit from them, as their bodies cannot process them. We call this resistance to therapy (RT).Because blood thinning is particularly important after operations people with RT may be at higher risk of their operation failing leading to amputation and/or problems such as heart attacks and strokes. Testing for RT has not traditionally been performed because it requires complex laboratory procedures. Recent development in technology now means that bedside tests are available for RT. We will use a simple beside test for RT in patients with severe PAD. We will use this test to see how many of these patients have RT and whether this affects their risk of complications after an operation. If we find that RT does affect outcomes for patients with PAD, the information obtained will be used to plan future research to determine if changing blood thinning therapy in people with CR improves their outcomes after surgery.

DETAILED DESCRIPTION:
Patients with peripheral arterial disease, a condition whereby arteries in the legs become narrow or blocked, are not only at a higher risk of limb loss but also of suffering heart attacks and strokes. To manage this risk and to ensure surgery for the blocked arteries is successful, they are prescribed tablets to make their blood less sticky, called antiplatelet agents. Aspirin and clopidogrel are the two tablets most commonly prescribed for this purpose.

In some patients, these two tablets are not effective as expected, because of interactions with other medications they are on or because their bodies cannot process them. This is known as resistance to antiplatelet therapy.

The main aim of this study is to establish how common resistance to aspirin and clopidogrel is in patients with peripheral arterial disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 years.
* Patients with severely symptomatic aorto-iliac and infra-inguinal peripheral arterial disease.
* Patients with the ability to provide written informed consent.
* Patients on antiplatelet therapy

Exclusion Criteria:

* Patients under the age of 18 years.
* Patients unable or unwilling to provide written informed consent.
* Patients with acute limb ischaemia of the lower limb.
* Patients with aneurysmal disease of the arteries of the lower limb.
* Patients with severe diabetic foot sepsis.
* Patients with a known history of clotting disorders
* Patients with inherited bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of interest is patients presenting electively or as an emergency with:
  * Disabling intermittent claudication (Rutherford stage III)
  * Ischaemic rest pain (Rutherford Stage IV)
  * Minor tissue loss due to peripheral arterial disease (Rutherford Stage V)
  * Ulceration or gangrene due to peripheral arterial disease (Rutherford Stage VI).
  Patients presenting with diabetic foot infection or diabetic foot sepsis will not be considered for
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To examine the feasibility of using the VerifyNow PRU and Aspirin assays to obtain estimates of the prevalence of resistance to antiplatelet therapy (aspirin & clopidogrel) in patients with symptomatic peripheral arterial disease. | 18 months
  Prevalence of resistance to aspirin and clopidogrel will be calculated as:
  Prevalence = (Number of patients resistant/Total study population) * 100
  Total estimated sample size of 150 participants.
  The VerifyNow PRU Test (CPT85576) is reported as P2Y12 Reaction Units (PRU). PRU measures the extent of platelet aggregation in the presence of a P2Y12 inhibitor.
  <180 PRU - suggests P2Y12 inhibitor effect 180-376 PRU - suggests lack of P2Y12 inhibitor effect.
  The VerifyNow Aspirin (CPT 85576) test is reported as Aspirin Reaction Units (ARU). ARU measures the extent of platelet aggregation in the presence of Arachidonic acid.
  </= 549 ARU - Evidence of platelet dysfunction due to aspirin > 550 ARU - No evidence of aspirin-induced platelet dysfunction.

SECONDARY OUTCOMES:
To examine whether resistance to antiplatelet therapy is associated with major adverse cardiac or limb events during the follow up interval of one year | 18 months
  Risk ratio = Cumulative incidence of major adverse cardiac/limb events in the Resistant Groups/Cumulative Incidence of Major events in the non-Resistant group
  Major adverse cardiac events = myocardial infarction, stroke, cardiovascular death Major adverse limb events = major amputation, acute limb ischaemia, re-operation
  Events will be assessed through interrogation of electronic medical records and phone calls with participants at both 6 months and one year follow up.
  Total estimated sample size of 150 participants.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Jane Messeder, MBChB, Principal Investigator — University of Leicester
Locations (1):
- University Hospitals Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No